CLINICAL TRIAL: NCT04242732
Title: Assessment of Patellar Stability in Patients Who Underwent Reconstruction of the Medium Patello-femoral Ligament With Fascia Lata Allograft: Comparison Between Conventional CT and Under Weight-bearing CT
Brief Title: Patellar Stability After MPFL Reconstruction With Fascia Lata Allograft: Conventional CT vs Under Weight-bearing CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CBCT-MPFL
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Patellofemoral Dislocation
Keywords: Patello femoral dislocation; Medial patello-femoral ligament; Sport trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MPFL reconstructed (Experimental): 20 patients with previous recurrent patella dislocation who underwent MPFL reconstruction surgery with fascia lata allograft between 2012 and 2013
  Interventions: Diagnostic Test: CT scan of the knee under weight-bearing with the Cone Beam Computed Tomography (CBCT) scanner system.; Diagnostic Test: Conventional CT scan

INTERVENTIONS:
Diagnostic Test: CT scan of the knee under weight-bearing with the Cone Beam Computed Tomography (CBCT) scanner system. — The patient will be evaluated under weight-bearing, with knee flexed at 30 ° and therefore with contracted thigh muscles. The measurement and maintenance of the 30 ° of flexion will be controlled by a goniometer applied laterally to the knee and fixed by means of an elastic band.
Diagnostic Test: Conventional CT scan — The patient will be evaluated in supine position, with the muscles relaxed and the knee in full extension by conventional CT scan

SUMMARY:
The objective of the present study is to compare the stability and alignment of the patella in patients with previous recurrent dislocation treated with medial patellar femoral ligament reconstruction with fascia lata allograft, 5 years after surgery by conventional CT and by CT under weight-bearing.

Conventional CT will be performed with the patient supine, the knee fully extended and with the muscles of the thigh and leg completely relaxed. On the same day, the patient will undergo a CT scan of the knee under weight-bearing with the Cone Beam Computed Tomography (CBCT) scanner system.

The CT images will be viewed through the PACS system by two independently expert radiologists who will measure the tilt, congruence angles and the TT-TG with the methodical notes described in the literature.

The use of a CT under weight-bearing allows for the first time to evaluate in a realistic way the stability and tracking of the patella, with the knee flexed and therefore with the activation of the quadriceps muscle.

DETAILED DESCRIPTION:
Patellofemoral disorders make up about 20% of all knee pathologies and are often a source of diagnostic and therapeutic doubts for the orthopedic surgeon. The incidence of patella dislocation is estimated to be 5.8 cases per 100,000 people, with values that become five times higher in patients aged between 10 and 17 years. Conservative treatment is preferable in the first case of acute dislocation, however the recurrence of this episode occurs in a percentage equal to 15 - 44% in these subjects.

Many surgical interventions have been described to correct the various factors that predispose to patellofemoral instability, with variable success rates (72% with the Hauser technique and 93% with the Roux-Goldthwait technique, 73% with that of Fielding and 78% with that of Trillat after a long follow-up.

The medial patello-femoral ligament (MPFL) is one of the main stabilizers of the patella in its movement on the femur; numerous studies have recently shown that this ligament is damaged in almost all cases, thus recognizing the role of the structure that most limits the patella in its lateral dislocation to the MPFL. Following these studies, the reconstruction of the MPFL as an elective treatment for relapsing patella dislocation has been recently proposed with countless surgical techniques that use various types of grafts: autologous tendons (the first in 1990 by Suganuma et al), tendons from donor (allograft) and synthetic ligaments.

Our team recently developed a minimally invasive MPFL reconstruction technique using an allograft tendon of the fascia lata with the aim of stabilizing the patella and limiting the patellofemoral arthritic degeneration in the medium to long term.

The imaging evaluation of instability and correct alignment of the patella, both in the pre-operative and in the post-surgery, is normally performed using magnetic resonance imaging or conventional CT. The CT offers the advantage of being able to make a very accurate morphological evaluation and therefore to be able to calculate with great precision the degrees of the tilt angle of the patella, the subluxation and the distance between the tibial tuberosity and the center of the trochlear sulcus (TT-TG ). The big limit of this method is that the patient is acquired supine, with the knee extended and with the muscles of the leg relaxed while it is well known how the knee flexion and the contraction of the quadriceps muscle possible in load, significantly affect the tracking of the patella on the trochlea. In literature, numerous studies show that the acquisition of the lying patient removes these determining factors (Callaghan; Draper; Tanaka) by altering the assessment of instability and malalignment. In a recent study by Marzo et al. it has been shown that in subjects suffering from instability of the patella, the evaluation under weight-bearing and with knee flexed by CT (CBCT Carestream) shows lower tilt angles, congruence and TT-TG than the evaluation in load and therefore the evaluation under load of the patellar alignment is more adequate to evaluate with precision these parameters.

The objective of the present study is to compare the stability and alignment of the patella in patients with previous relapsing dislocation treated with reconstruction surgery by means of a medial patellar ligament with lata band allograft 5 years after surgery by conventional CT and by CT under weight-bearing.

The assessments are carried out in a group of 20 patients with previous recurrent patella dislocation who underwent reconstruction surgery between 2012 and 2013 via a medial patello-femoral ligament with fascia lata allograft at the Orthopedic and Traumatologic Clinic 2nd of the Rizzoli Orthopedic Institute. The patients will be contacted by phone and a follow-up visit will be scheduled which is normally carried out 5 years after the operation to evaluate the stability of the patella and therefore the patient's clinical condition. The patient will undergo a clinical examination and radiological control with conventional CT at the Rizzoli Orthopedic Institute. Conventional CT will be performed with the patient supine, the knee fully extended and with the muscles of the thigh and leg completely relaxed. On the same day, the patient will undergo a CT scan of the knee under weight-bearing with the Cone Beam Computed Tomography (CBCT) scanner system.The CT images will be viewed through the PACS system by two independently expert radiologists who will measure the tilt, congruence angles and the TT-TG with the methodical notes described in the literature.

The use of a CT under weight-bearing allows for the first time to evaluate in a realistic way the stability and tracking of the patella, with the knee flexed and therefore with the activation of the quadriceps muscle.

ELIGIBILITY:
Inclusion Criteria:

* Who is able to provide informed consent and who agrees to sign the Informed Consent Form approved by the Ethics Committee (EC).
* Subject who underwent reconstruction of the MPFL using a minimally invasive technique using a fascia fascia allograft, performed at the Rizzoli Orthopedic Institute between 2012 and 2013 by the team of Prof. Zaffagnini.

Exclusion Criteria:

* patients with severe morphostructural deformities or other pathologies affecting the knee and lower limb
* patients with serious systemic vascular and neurological pathologies
* patients unable to perform a CT scan under weight-bearing
* State of pregnancy.
* Obese or with body mass index BMI> 30 kg / m2.
* Association of Trocleoplasty (intervention that produces degenerative changes of the joint in high percentage)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-05-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Patellar Tilt Angle | 24 months
  The tilt angle is defined as the angle subtended by a line joining the medial and lateral edges of the patella and the horizontal plane on the axial plane, measured both by conventional CT scan with the knee extended and by CT scan under weight bearing conditions with the knee flexed at 30°.
Patellar Congruence Angle | 24 months
  Angle made by a line parallel to the posterior condyles and the line joining the edges of the patella on the axial plane, measured under weight-bearing with knee flexed at 30° and supine with knee extended.
Tibial tuberosity-trochlear groove distance | 24 months
  Radiographic parameter measured by CT scan both under weight-bearing with knee flexed at 30° and supine with knee extended.

CONTACTS AND LOCATIONS:
Overall Officials: Giada Lullini, MD, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arnbjornsson A, Egund N, Rydling O, Stockerup R, Ryd L. The natural history of recurrent dislocation of the patella. Long-term results of conservative and operative treatment. J Bone Joint Surg Br. 1992 Jan;74(1):140-2. doi: 10.1302/0301-620X.74B1.1732244.
- [Result] Chrisman OD, Snook GA, Wilson TC. A long-term prospective study of the Hauser and Roux-Goldthwait procedures for recurrent patellar dislocation. Clin Orthop Relat Res. 1979 Oct;(144):27-30. PMID 535237
- [Result] Crosby EB, Insall J. Recurrent dislocation of the patella. Relation of treatment to osteoarthritis. J Bone Joint Surg Am. 1976 Jan;58(1):9-13. PMID 1249117
- [Result] Dejour H, Walch G, Neyret P, Adeleine P. [Dysplasia of the femoral trochlea]. Rev Chir Orthop Reparatrice Appar Mot. 1990;76(1):45-54. French. PMID 2140459
- [Result] Desio SM, Burks RT, Bachus KN. Soft tissue restraints to lateral patellar translation in the human knee. Am J Sports Med. 1998 Jan-Feb;26(1):59-65. doi: 10.1177/03635465980260012701. PMID 9474403
- [Result] Fielding JW, Liebler WA, Krishne Urs ND, Wilson SA, Puglisi AS. Tibial tubercle transfer: a long-range follow-up study. Clin Orthop Relat Res. 1979 Oct;(144):43-4. PMID 535248
- [Result] Hautamaa PV, Fithian DC, Kaufman KR, Daniel DM, Pohlmeyer AM. Medial soft tissue restraints in lateral patellar instability and repair. Clin Orthop Relat Res. 1998 Apr;(349):174-82. doi: 10.1097/00003086-199804000-00021. PMID 9584380
- [Result] Hefti F, Muller W, Jakob RP, Staubli HU. Evaluation of knee ligament injuries with the IKDC form. Knee Surg Sports Traumatol Arthrosc. 1993;1(3-4):226-34. doi: 10.1007/BF01560215. PMID 8536037
- [Result] Iwano T, Kurosawa H, Tokuyama H, Hoshikawa Y. Roentgenographic and clinical findings of patellofemoral osteoarthrosis. With special reference to its relationship to femorotibial osteoarthrosis and etiologic factors. Clin Orthop Relat Res. 1990 Mar;(252):190-7. PMID 2302884
- [Result] Kodraliu G, Mosconi P, Groth N, Carmosino G, Perilli A, Gianicolo EA, Rossi C, Apolone G. Subjective health status assessment: evaluation of the Italian version of the SF-12 Health Survey. Results from the MiOS Project. J Epidemiol Biostat. 2001;6(3):305-16. doi: 10.1080/135952201317080715. PMID 11437095
- [Result] Kujala UM, Jaakkola LH, Koskinen SK, Taimela S, Hurme M, Nelimarkka O. Scoring of patellofemoral disorders. Arthroscopy. 1993;9(2):159-63. doi: 10.1016/s0749-8063(05)80366-4. PMID 8461073
- [Result] Zaffagnini S, Grassi A, Marcheggiani Muccioli GM, Luetzow WF, Vaccari V, Benzi A, Marcacci M. Medial patellotibial ligament (MPTL) reconstruction for patellar instability. Knee Surg Sports Traumatol Arthrosc. 2014 Oct;22(10):2491-8. doi: 10.1007/s00167-013-2751-1. Epub 2013 Nov 7. PMID 24196574
- [Result] Marcacci M, Zaffagnini S, Iacono F, Visani A, Petitto A, Neri NP. Results in the treatment of recurrent dislocation of the patella after 30 years' follow-up. Knee Surg Sports Traumatol Arthrosc. 1995;3(3):163-6. doi: 10.1007/BF01565476. PMID 8821272
- [Result] Monticone M, Ferrante S, Salvaderi S, Rocca B, Totti V, Foti C, Roi GS. Development of the Italian version of the knee injury and osteoarthritis outcome score for patients with knee injuries: cross-cultural adaptation, dimensionality, reliability, and validity. Osteoarthritis Cartilage. 2012 Apr;20(4):330-5. doi: 10.1016/j.joca.2012.01.001. Epub 2012 Jan 10. PMID 22285738
- [Result] Outerbridge RE. The etiology of chondromalacia patellae. 1961. Clin Orthop Relat Res. 2001 Aug;(389):5-8. doi: 10.1097/00003086-200108000-00002. No abstract available. PMID 11501822
- [Result] Smith TO, Walker J, Russell N. Outcomes of medial patellofemoral ligament reconstruction for patellar instability: a systematic review. Knee Surg Sports Traumatol Arthrosc. 2007 Nov;15(11):1301-14. doi: 10.1007/s00167-007-0390-0. Epub 2007 Aug 8. PMID 17684729
- [Result] Tegner Y, Lysholm J. Rating systems in the evaluation of knee ligament injuries. Clin Orthop Relat Res. 1985 Sep;(198):43-9. PMID 4028566
- [Result] TRILLAT A, DEJOUR H, COUETTE A. [DIAGNOSIS AND TREATMENT OF RECURRENT DISLOCATIONS OF THE PATELLA]. Rev Chir Orthop Reparatrice Appar Mot. 1964 Nov-Dec;50:813-24. No abstract available. French. PMID 14256559
- [Result] Zaffagnini S, Colle F, Lopomo N, Sharma B, Bignozzi S, Dejour D, Marcacci M. The influence of medial patellofemoral ligament on patellofemoral joint kinematics and patellar stability. Knee Surg Sports Traumatol Arthrosc. 2013 Sep;21(9):2164-71. doi: 10.1007/s00167-012-2307-9. Epub 2012 Nov 24. PMID 23179455
- [Result] Zaffagnini S, Marcheggiani Muccioli GM, Grassi A, Bonanzinga T, Marcacci M. Minimally invasive medial patellofemoral ligament reconstruction with fascia lata allograft: surgical technique. Knee Surg Sports Traumatol Arthrosc. 2014 Oct;22(10):2426-30. doi: 10.1007/s00167-014-2940-6. Epub 2014 Mar 22. PMID 24658149
- [Result] Marzo J, Kluczynski M, Notino A, Bisson L. Comparison of a Novel Weightbearing Cone Beam Computed Tomography Scanner Versus a Conventional Computed Tomography Scanner for Measuring Patellar Instability. Orthop J Sports Med. 2016 Dec 7;4(12):2325967116673560. doi: 10.1177/2325967116673560. eCollection 2016 Dec. PMID 28050572